CLINICAL TRIAL: NCT02582528
Title: Pilot Study of Cognitive Remediation and Motivational Interviewing on Cognition and Functioning in Young People at Risk of Serious Mental Illness
Brief Title: Cognitive Remediation in Youth at Risk of Serious Mental Illness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Danijela Piskulic, Research Fellow, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCalgary-MAT
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Depression; Psychosis; Anxiety; Mental Illness
Keywords: cognitive remediation; cognition; youth; mental health; functional outcome
MeSH Terms: conditions — Depression; Psychotic Disorders; Anxiety Disorders; Mental Disorders; Psychological Well-Being | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cognitive remediation treatment and MI (Experimental): Cognitive remediation treatment consisting of a novel computerized training called My Brain Solutions (MBS) and motivational interviewing, a client-centered, directive method for enhancing intrinsic motivation to change.
  Interventions: Behavioral: Cognitive remediation treatment; Behavioral: Motivational Interviewing
- cognitive remediation treatment (Active Comparator): Cognitive remediation treatment consisting of a novel computerized training called My Brain Solutions (MBS)
  Interventions: Behavioral: Cognitive remediation treatment

INTERVENTIONS:
Behavioral: Cognitive remediation treatment — Cognitive remediation treatment consisting of a novel computerized training called My Brain Solutions (MBS)
  Other Names: My Brain Solutions
Behavioral: Motivational Interviewing — A client-centered, directive method for enhancing intrinsic motivation to change.
  Other Names: MI
  Arms: cognitive remediation treatment and MI

SUMMARY:
The primary aim of the project is to test the effectiveness of a cognitive remediation treatment (CRT) program, My Brain Solutions (MBS), in addition to motivational interviewing (MI) in improving cognition and functional outcome of individuals at risk of SMI. An active control treatment consisting of CRT alone will be used. Hypotheses: 1. Both study groups will have improvement in cognition at the end of treatment; 2. CRT+MI group will have increased treatment adherence and superior improvements in cognition at the end of treatment and 12 months post baseline compared to the CRT only group; Secondary Hypothesis: 3. Improved cognition will be associated with improved functional outcome.

DETAILED DESCRIPTION:
Individuals identified to be at clinical high risk of psychosis (CHR) of psychosis already evidence cognitive deficits, which increase around the time of conversion. Much less is known about individuals that may be at risk of other serious mental disorders (SMI). However, early reports are suggesting that young people at risk of SMI who are deemed to have "attenuated syndromes" according to the clinical staging model of mental health disorders already evidence cognitive deficits. Therefore, cognition is an excellent treatment target. Furthermore, there is clear evidence, in both established psychiatric disorders such as schizophrenia, depression and bipolar disorder, and in CHR samples, that deficits in cognition are associated to poor functional outcome. Thus, treatments targeting cognition may consequently improve functional outcome. This is a pilot project to determine feasibility and sample size for a large randomized controlled trial of cognitive remediation therapy (CRT) in people at risk of SMI with CIHR and AIHS funding targets. The primary aim of the project is to test the effectiveness of a novel computerized CRT program in improving cognition in youth at risk of SMI following the addition of a counseling intervention, MI, to improve adherence to CRT. One group will receive CRT and the other CRT plus MI. Hypotheses: 1. Both study groups will have improvement in cognition at the end of treatment; 2. CRT+MI group will have increased treatment adherence and superior improvements in cognition at the end of treatment and 12 months post baseline compared to the CRT only group; Secondary Hypothesis: 3. Improved cognition will be associated with improved functional outcome. This is a longitudinal, single blind, controlled pilot trial of CRT in persons at risk of SMI. Twenty-eight participants will be recruited from the Adolescent Mental Health: Canadian Psychiatric Risk and Outcome Study (PROCAN) study at the Calgary site led by Dr. J. Addington. Participants in the PROCAN project who meet operationally defined criteria as being at risk of SMI by meeting attenuated syndromes criteria will be included. Participants will be randomized to either the CRT condition consisting of a novel program called My Brain Fitness (MBS) and motivational interviewing (MI) or a control condition consisting of CRT alone, and will receive training that will be administered over a period of 10 weeks. Assessments will occur at baseline, post treatment (3 months) and at 12 months after baseline. Half of all participants will receive individual 1 hr MI once every 2 weeks for the duration of the cognitive remediation component of the study. The study clinicians who are master level psychologists, will deliver MI ensuring engagement of study participants. Time spent in therapy will be monitored and recorded. All of the data necessary for this study will be collected as part of the PROCAN assessment at baseline and 12 months. The one exception is that we will do an assessment of cognitive function, clinical symptoms and functional outcome at 10 weeks or immediately post treatment, which will take approximately 2.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 14-25 years with subthreshold mood and psychotic symptoms.

Exclusion Criteria:

* (i) meet criteria for current or lifetime Axis I bipolar or psychotic disorder (other Axis I disorders will not be exclusionary as they may be precursors to mood or psychotic disorders);
* (ii) IQ < 70;
* (iii) past or current history of a significant central nervous system disorder or serious medical disorder; and
* (iv) current pharmacological treatment that would be considered as an adequate trial of treatment for a SMI.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Cognitive function assessment pre- and post-CRT in youth at risk of SMI using WebNeuro computerized cognitive battery | one year
  A web-based battery for assessing general and emotional cognition, completed at any computer using mouse and keyboard. The assessment has been validated against traditional paper-and-pencil tests and with established reliability, cross-cultural consistency and norms.

SECONDARY OUTCOMES:
Social functioning assessment pre- and post-CRT in youth at risk of SMI using Global Functioning: Social (GFS) scale. | one year
  GFS consists of 10 items that are used to provide a rating of current social functioning. Scores range between 1 and 10, with 10 indicating superior functioning and 1 representing severe dysfunction.
Social functioning assessment pre- and post-CRT in youth at risk of SMI using Global Functioning: Role (GFR) scale. | one year
  GFR consists of 10 items that are used to provide a rating of current role or occupational functioning. Scores range between 1 and 10, with 10 indicating superior functioning and 1 representing severe dysfunction.
Functional capacity assessment pre- and post-CRT in youth at risk of SMI using Social Skills Performance Assessment (SSPA). | one year
  The SSPA is focused on both verbal and nonverbal social skills that are needed to succeed in two different social interaction tasks. Higher scores on the SSPA indicate better social skills.

CONTACTS AND LOCATIONS:
Overall Officials: Danijela Piskulic, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided